CLINICAL TRIAL: NCT01474525
Title: Managing Diabetes During Pregnancy in the Wireless Age: a RCT of Glucose Telemonitoring
Brief Title: Managing Diabetes During Pregnancy in the Wireless Age
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Collaborators: Ontario Ministry of Health and Long Term Care (Other Government)
Responsible Party: Principal Investigator, Alexander Gordon Logan, Principal Investigator, Samuel Lunenfeld Research Institute, Mount Sinai Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AFP6075
Record Dates: First submitted 2011-07-20; First posted 2011-11-18 (Estimated); Last update posted 2011-11-21 (Estimated); Status verified 2011-11

CONDITIONS: Gestational Diabetes Mellitus; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes, Gestational; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Telemonitoring (Experimental)
  Interventions: Device: Home Blood Glucose Telemonitoring System
- Usual Care (Active Comparator)
  Interventions: Device: Home Blood Glucose Telemonitoring System

INTERVENTIONS:
Device: Home Blood Glucose Telemonitoring System — The system is designed to send the measured blood glucose values directly to a hospital server. Values recorded by the glucometer are sent to the Blackberry® cell phone. A special removable Bluetooth® adapter unit is required for data transmission from the glucometer to the Blackberry®. The patient must then select on the Blackberry® the meal period the last measurement corresponds. The cellular phone serves as the platform for data-transmission to the central server. The threshold number of readings can be set for each patient individually through the web-interface. The system can be accessed by both the patients and the care providers through a secure web-interface.
  Apart from collecting values the system generates automated adherence reminders to patients and high/low blood glucose alert messages to both patients and their care providers.

SUMMARY:
This Randomized Controlled Trial (RCT) will test the efficacy of a home blood glucose telemonitoring system against usual care in women with gestational diabetes mellitus (GDM) or type 2 diabetes mellitus (T2DM) during pregnancy. We hypothesize that the system can improve glycemic control in patients, assessed using the mean blood glucose during gestation as the primary outcome measure.

DETAILED DESCRIPTION:
Establishing good glycemic control is crucial for the treatment of patients with gestational diabetes mellitus (GDM) and type 2 diabetes mellitus (DM2). High levels of blood glucose in pregnancy may lead to complications during delivery and pose threat to the fetus. The self-monitoring of blood glucose (SMBG) by patients at home is used to provide clinicians with information to make adjustments to treatment plans. Patients record the values and present them at their next meeting with the physician. As such, SMBG by the patients is an important part of disease management and a method for clinicians to follow a patient's day-to-day response to a treatment regime.

The system is designed to send the blood glucose values from the patients' glucometers wirelessly to the server where they can be viewed by the patients' health care providers. The system generates automated adherence reminders to patients and alert messages to both patients and their care providers. The system will provide clinicians with better access to the patient data, so that they may better manage their case loads, make timely clinical decisions, and ultimately provide better patient care.

ELIGIBILITY:
Inclusion Criteria:

* patients must be pregnant
* diagnosed with gestational diabetes or Type 2 diabetes
* must be comfortable with instructions in English and be able to express themselves using simple phrases in English.

Exclusion Criteria:

* unable to complete self monitoring of blood glucose (SMBG) for any reason
* uncomfortable with the use of the telemonitoring equipment
* develop an acute illness requiring hospitalization, where they may deviate from the normal delivery of care
* refusal to sign consent form or to carry out the demands made by the study

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-01; Primary Completion 2012-03 (Estimated); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
Mean blood glucose, based on the highest post-prandial blood glucose reading for each day, by trimester | from the baseline to the delivery date
  An average of 12 weeks.

SECONDARY OUTCOMES:
Mean fasting and post-prandial blood glucose by trimester | from the baseline to the delivery date
  An average of 12 weeks.
Percentage of values within recommended guidelines | from the baseline to the delivery date
  An average of 12 weeks.
Adherence: Percentage of values recorded over expected number of values | from the baseline to the delivery date
  An average of 12 weeks.
Adherence: Average number of values per day | from the baseline to the delivery date
  An average of 12 weeks.
Onset of labour and mode of delivery | at exit (delivery)
  An average of 3 days.
Fetal outcomes: gestational age at delivery, birth weight (by gender), percentage of macrosomia, large for gestational age (LGA) and small for gestational age (SGA), APGAR at 1 and 5 minutes | at exit (delivery)
  An average of 1 day.
Perinatal complications (i.e. premature, NICU admission, jaundice, shoulder dystocia, hypoglycemia) | at exit (delivery)
  An average of 1 week.
Provider usage: number of logins onto the system, average amount of time spent on the system per week | for the duration of the study
  An average of 12 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander G Logan, MD, FRCP(C), Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Leadership Sinai Centre for Diabetes, Toronto, Ontario, Canada

REFERENCES:
- [Background] HAPO Study Cooperative Research Group; Metzger BE, Lowe LP, Dyer AR, Trimble ER, Chaovarindr U, Coustan DR, Hadden DR, McCance DR, Hod M, McIntyre HD, Oats JJ, Persson B, Rogers MS, Sacks DA. Hyperglycemia and adverse pregnancy outcomes. N Engl J Med. 2008 May 8;358(19):1991-2002. doi: 10.1056/NEJMoa0707943. PMID 18463375
- [Background] Crowther CA, Hiller JE, Moss JR, McPhee AJ, Jeffries WS, Robinson JS; Australian Carbohydrate Intolerance Study in Pregnant Women (ACHOIS) Trial Group. Effect of treatment of gestational diabetes mellitus on pregnancy outcomes. N Engl J Med. 2005 Jun 16;352(24):2477-86. doi: 10.1056/NEJMoa042973. Epub 2005 Jun 12. PMID 15951574
- [Background] Feig DS, Palda VA. Type 2 diabetes in pregnancy: a growing concern. Lancet. 2002 May 11;359(9318):1690-2. doi: 10.1016/S0140-6736(02)08599-9. No abstract available. PMID 12020549
- [Background] Langer O. Type 2 diabetes in pregnancy: exposing deceptive appearances. J Matern Fetal Neonatal Med. 2008 Mar;21(3):181-9. doi: 10.1080/14767050801929497. PMID 18297573
- [Background] Kinsley B. Achieving better outcomes in pregnancies complicated by type 1 and type 2 diabetes mellitus. Clin Ther. 2007;29 Suppl D:S153-60. doi: 10.1016/j.clinthera.2007.12.015. PMID 18191067
- [Background] Yang J, Cummings EA, O'connell C, Jangaard K. Fetal and neonatal outcomes of diabetic pregnancies. Obstet Gynecol. 2006 Sep;108(3 Pt 1):644-50. doi: 10.1097/01.AOG.0000231688.08263.47. PMID 16946226